CLINICAL TRIAL: NCT04405817
Title: Outcome of Patients Treated With Extracorporeal Life Support
Brief Title: Outcome of Patients Treated With ECLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Department of Cardiac Surgery, Nanjing Medical University
Other Study IDs: ECLS-Jsph
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Cardiogenic Shock; Cardiac Arrest; Heart Failure; Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest; Heart Failure; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECMO — ECMO for circulatory and/or respiratory support

SUMMARY:
Extracorporeal life support (ECLS), also called extracorporeal membrane oxygenation (ECMO), is an extracorporeal technique of providing effective circulatory and (or) respiratory failure, with a growing number of critically ill patients benefit from it. The aim of this study is to investigate the outcome of patients treated With ECMO, and to evaluate the short-term and long-term outcomes of patients with ECLS.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ECMO for circulatory and/or respiratory support

Exclusion Criteria:

* Refusal of consent

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving ECMO for circulatory and/or respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of death from any cause, resuscitated circulatory arrest, and implantation of another mechanical circulatory support device | 30 days after ECMO implantation

SECONDARY OUTCOMES:
All-cause mortality | 30 days after ECMO implantation
All-cause mortality | 12 months after ECMO implantation

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided